CLINICAL TRIAL: NCT04579874
Title: Clinical Performance Evaluation of LIVERFASt Tests to Determine Fibrosis Staging, Inflammatory Activity and Steatosis Grading Compared w/ Liver Biopsy in Patients w/ Metabolic Factors & Presumed Non-Alcoholic Fatty Liver Disease (NAFLD).
Brief Title: Clinical Performance of LIVERFASt Test Compared w/ Liver Biopsy in Patients w/ NAFLD.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fibronostics USA, Inc (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Fibro-US-001-0200
Record Dates: First submitted 2020-09-25; First posted 2020-10-08 (Actual); Last update posted 2022-08-02 (Actual); Status verified 2022-07

CONDITIONS: Non-Alcoholic Fatty Liver Disease; Non-Alcoholic Steatohepatitis; Liver Fibroses; Liver Inflammation; Liver Steatoses
Keywords: LIVERFASt; Liver biopsy; Liver Fibrosis; Liver Activity; Liver Steatosis; Non-invasive serum biomarker; Neural Network; Artificial Intelligence Machine Learning; Algorithm based test
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Liver Cirrhosis; Hepatitis; Fatty Liver

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- LIVERFASt validation (Experimental): blood draw for LIVERFASt
  Interventions: Diagnostic Test: LIVERFASt

INTERVENTIONS:
Diagnostic Test: LIVERFASt — blood draw

SUMMARY:
The primary objective of this study is to assess the clinical performance of LIVERFAStTM In Vitro Diagnostic (IVD) Tests (Fibrosis score, Activity score and Steatosis score) in NAFLD suspected patients for staging of fibrosis and for grading of inflammatory activity and steatosis, taking as reference the liver biopsy with histological classification of the elementary lesions determined according to SAF scores (Bedossa P., Hepatology 2012).

The secondary objective is to assess the performance of LIVERFAStTM for the histological definition of NAFLD, including NAFL and NASH and severe NASH

DETAILED DESCRIPTION:
Chronic liver diseases (CLDs), such as chronic viral hepatitis, nonalcoholic fatty liver diseases (NAFLD) and nonalcoholic steatohepatitis (NASH), are a leading cause of morbidity and mortality globally and usually develops over many years. The prevalence of NAFLD has increased in recent years (15% in 2005 to 25% in 2010) mainly due to the increase prevalence of obesity and diabetes. As, approximately 20% of NAFLD cases develop NASH, the associated increase in NASH during the same period is to be expected (33% in 2005 to 59.1% in 2010).

As a result, staging of liver fibrosis is essential in determining the prognosis and optimal treatment for patients with NASH. Furthermore, evaluation of fibrosis in NAFLD patients can help refine treatment options designed to prevent the progression to NASH.

One recent study demonstrates significant sampling variability of routine liver biopsy in patients with NAFLD (Ratziu V. et al. Gastroenterology 2008). The diagnosis of NASH would have been missed in 35% and the discordance for steatosis grading was encountered in 22% of patients.

Developing safe and easily accessible noninvasive modalities to accurately evaluate fibrosis stage of NAFLD and NASH is of utmost importance in clinical practice.

Fibronostics breaks through the burden to serve patients. By empowering their providers with IVD clinical tools within the clinic, the ability to ensure screening and clinical adherence is assured, and the ease for early detection profoundly shifts the $2B economic burden.

LIVERFASt is a non-invasive clinical and staging In-Vitro-Diagnostic (IVD) tool, which has been developed as an alternative to liver biopsy. LIVERFASt is a safe, and reproducible tool which provides surrogate grading and staging of the three elementary features of NASH: steatosis, inflammatory activity and fibrosis.

LIVERFAStTM combines age, gender, weight and height with common liver function tests (ALT, AST, GGT, total bilirubin), lipid profile (total cholesterol, triglycerides), fasting glucose and three specific proteins of the liver with hepatoprotective functions and predictive value in NAFLD -alpha2-macroglobulin (A2M), haptoglobin (HAP) and apolipoprotein A1 (APOA1).

The main aim of this study is to evaluate the clinical value of LIVERFAStTM as a non-invasive biopsy-proven surrogate assessment of non-alcoholic fatty liver disease.

This is a cohort cross-sectional prospective, multi-centre study of an algorithm-based assessment of liver fibrosis, inflammatory activity (steatohepatitis) and steatosis compared to the histological assessment provided by liver biopsy performed in patients with suspected non-alcoholic steatohepatitis (NASH).

ELIGIBILITY:
Inclusion Criteria:

* • Consenting patients with suspected NAFLD (by any means) having had undergone liver biopsy as part as their routine management, simultaneously or within six months from the day of blood sampling for LIVERFAStTM test.

  * Aged 18 to 80 years old, inclusive
  * Male or Female from any ethnicity
  * Willing to undergo blood sampling for LIVERFAStTM testing after 6 to 12 hours fasting
  * Willing to allow histological lecture by a pathologist for NASH-CRN and SAF scoring systems analysis of the liver biopsy
  * Willing and able to allow access to requested data and who were informed and signed the consent form.

Exclusion Criteria:

* • Inability to provide informed consent

  * Patients who may be uncooperative with the sample collection procedures
  * History of known Severe coagulopathy
  * History of known Hepatic abscess
  * Renal failure undergoing dialysis (GFR<45)
  * History of Malignancy in the past 2 years
  * Previous liver transplantation
  * Suffering with a terminal illness or any other conditions or diseases that the investigator considers inappropriate for study participation
  * Secondary causes of hepatic fat accumulation such as significant alcohol consumption, long-term use of a steatogenic medication, ()
  * Ongoing or recent significant alcohol consumption defined as >21 standard drinks on average per week in men and >14 standard drinks on average per week in women.8 Approximately 10 g of alcohol equals one 'drink' unit. One unit equals 1 ounce of distilled spirits, one 12-oz beer, or one 4-oz glass of wine.
  * Total parenteral nutrition within 3 months of interview
  * Short bowel syndrome
  * History of gastric or jejunoileal bypass preceding the diagnosis of NAFLD. Bariatric surgery performed concomitant with or following the diagnosis of NAFLD does not exclude enrollment of patients.
  * History of biliopancreatic diversion
  * Evidence of advanced liver disease defined as a Child-Pugh-Turcotte score of equal to or greater than 10
  * Evidence of chronic hepatitis B as marked by the presence of HBsAg in serum (patients with isolated antibody to hepatitis B core antigen, anti-HBc, are not excluded)
  * Evidence of chronic hepatitis C as marked by the presence of anti-HCV and HCV RNA in serum; patients with anti-HCV with PCR negative should not be excluded
  * Low alpha-1-antitrypsin level and ZZ phenotype (both determined at the discretion of the investigator)
  * History of Wilson's disease
  * Known glycogen storage disease
  * Known dysbetalipoproteinemia
  * Known phenotypic hemochromatosis (determined at the discretion of the investigator)
  * History of primary biliary cholangitis (PBC)/primary biliary sclerosis (PSC)
  * Hepatic vascular lesions (determined at the discretion of the investigator)
  * History of liver liver granulomas sarcoidosis, and infectious diseases such as tuberculosis)
  * Congenital hepatic fibrosis, polycystic liver disease
  * Other metabolic/congenital liver disease
  * Evidence of systemic infectious disease
  * Known HIV positive
  * Disseminated or advanced extrahepatic malignancy
  * Conditions that could interfere with LIVERFASt parameters and could lead to risk of false positive/ false negative results:

    1. Drug induced liver-injury (DILI), acute alcoholic hepatitis
    2. Acute inflammatory syndrome or sepsis Active drug use or dependence that, in the opinion of the study investigator, would interfere with adherence to study requirements

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 241 (Actual)
Dates: Start 2021-01-07 (Actual); Primary Completion 2021-12-15 (Actual); Study Completion 2022-04-15 (Actual)

PRIMARY OUTCOMES:
Clinical performance of LIVERFASt Tests to determine liver fibrosis scores and staging compared with Liver Biopsy in patients with presumed Non-Alcoholic Fatty Liver Disease (NAFLD). | 12 months
  Primary:
  Clinical performance of the LIVERFASt Fibrosis score using the results of five serum biomarkers (A2M, Haptoglobin, ApoA1, Total Bilrubin and GGT) for the over-all diagnostic of liver fibrosis (F0, F1, F2, F3 and F4 stages) using Binary and Non-Binary-Area Under the ROC curve
Clinical performance of LIVERFASt Tests to determine inflammatory activity scores and staging compared with Liver Biopsy in patients with presumed Non-Alcoholic Fatty Liver Disease (NAFLD). | 12 months
  Clinical performance of the LIVERFASt Activity scores using the results of six serum biomarkers (A2M, Haptoglobin, ApoA1, Total Bilrubin, GGT and ALT) for the over-all diagnostic of inflammatory activity (A0, A1, A2, A3 and A4 grades) using Binary and Non-Binary-Area Under the ROC curve
Clinical performance of LIVERFAStTM Tests to determine steatosis grading compared with Liver Biopsy in patients with presumed Non-Alcoholic Fatty Liver Disease (NAFLD). | 12 months
  Clinical performance of the LIVERFAstTM Steatosis grading tests using the results of ten serum biomarkers (A2M, Haptoglobin, ApoA1, Total Bilrubin, GGT, ALT, AST, Triglyceride, Cholesterol and Fasting Blood Glucose) for the over-all diagnostic of steatosis (S0, S1, S2 and S3), using Binary and Non-Binary-Area Under the ROC curve

SECONDARY OUTCOMES:
Clinical performance evaluation of the LIVERFASt Tests to evaluate and measure the definition of NAFLD based on fibrosis staging (F0, F1, F2, F3 and F4), inflammatory activity (A0, A1, A2, A3 and A4) and steatosis grading (S0, S1, S2, and S3). | 12 months
  Secondary
  200 adult men and women who are between the ages of 18-80 years old patients who have undergone liver biopsy with suspected non-alcoholic fatty liver disease within six (6) months of the enrollment and have undergone blood sampling for LIVERFASt testing using the generated results of ten serum biomarkers, namely: A2M, Haptoglobin, ApoA1, Total Bilrubin, GGT, ALT, AST, Triglyceride, Cholesterol and Fasting Blood Glucose, for the over-all diagnosis of fibrosis (F0, F1 to F4), activity (A0, A1 to A4) and steatosis (S0, S1 to S3). Performance (Bin-AUROC) of the LIVERFASt using the results of the combination of the ten biomarkers for the NAFLD definitions of NAFL, NASH and significant NASH (>S1≥A2≥F2)

CONTACTS AND LOCATIONS:
Overall Officials: Ronald Quiambao, MD, Study Director — Fibronostics USA, Inc; Imtiaz Alam, MD, Principal Investigator — Ohio Gastroenterology and Liver Institute; Sven Henrichwark, Study Chair — Fibronostics USA, Inc
Locations (8):
- United States (8):
  - Henry Ford Health System, Detroit, Michigan
  - St. Louis University, St Louis, Missouri
  - Northwell Health, Inc, Manhasset, New York
  - GCGA Physicians, LLC, Cincinnati, Ohio
  - Methodist Health System Clinical Research Institute, Dallas, Texas
  - Baylor College of Medicine, Houston, Texas
  - Houston Methodist Research Institute, Houston, Texas
  - Liver Associates of Texas, P.A., Houston, Texas